CLINICAL TRIAL: NCT02582957
Title: Sigh Ventilation to Increase Ventilator-Free Days in Victims of Trauma at Risk for Acute Respiratory Distress Syndrome
Acronym: SiVent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1512M81688
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Shock Lung; Acute Chest Syndrome; Respiratory Distress Syndrome, Adult; Respiratory insufficiency; Trauma
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Chest Syndrome; Respiratory Insufficiency; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sigh breaths (Experimental): Sigh breaths consisting of a Tidal volume (VT) that produces a plateau pressure (Pplat) of 35 cmH2O (or 40 cmH2O in patients with BMIs > 35 or in patients with moderate or severe abdominal distension from ascites, blood and/or ileum, or prone patients). The sigh breaths will be delivered once every 6 minutes, as part of usual invasive mechanical ventilation.
  Interventions: Other: Sigh breaths
- Usual Care (No Intervention): Usual care, meaning that the treating physician will be free to treat the patient in any way he or she sees fit, including utilizing invasive mechanical ventilation as they wish.

INTERVENTIONS:
Other: Sigh breaths — Sigh breaths delivered once every 6 minutes, as part of usual invasive mechanical ventilation.
  Arms: Sigh breaths

SUMMARY:
A randomized, concurrent controlled trial to assess if adding sigh breaths to usual invasive mechanical ventilation of victims of trauma who are at risk of developing ARDS will decrease the number of days they require invasive mechanical ventilation.

DETAILED DESCRIPTION:
Patients in intensive care units (ICUs) as a result of injuries resulting from penetrating or non-penetrating trauma who are intubated and receiving invasive mechanical ventilation will be randomized to either usual care or usual care with the addition of sigh breaths given once every 6 minutes. Patients will be randomized to one of the two study arms as soon as possible, but not longer than 24 hours after initiation of invasive mechanical ventilation. Patients will be followed for 28 days to assess ventilator-free days (VFDs), mortality, ICU-free days, and the occurrence of complications.

ELIGIBILITY:
Inclusion Criteria:

Patients in an intensive care unit (ICU) as a result of injuries resulting from penetrating or non-penetrating trauma who are intubated and receiving invasive mechanical ventilation who also have one or more of the following:

1. Traumatic brain injury
2. > 1 long bone fractures
3. Shock on arrival in the Emergency Department (systolic BP < 90 mmHg)
4. Lung contusion
5. Receipt of > 6 units of blood

Exclusion Criteria:

1. Inability to obtain consent from the patient or his/her legally authorized representative (LAR)
2. Unwillingness of the treating physician to use sigh ventilation as all treating physicians must have equipoise with respect to the intervention
3. Age limitations per Institutional Review Board regulations
4. Undergoing invasive mechanical ventilation for > 24 hours, excluding any time during which the patient was being ventilated in the operating room, CT or IR, as this could represent too long a delay in instituting the intervention for it to have a chance of being effective
5. Presence of malignancy or other irreversible disease or condition for which the six month mortality is estimated to exceed 50% (e.g., chronic liver disease with a Child-Pugh Score of 10-15, malignancy refractory to treatment) as this could affect the clinical course and cloud interpretation of the endpoints
6. Women who are pregnant (negative pregnancy tests required on women of child-bearing age) per Human Subjects regulations
7. Prisoners, per Human Subjects regulations
8. Neurological condition that could impair spontaneous ventilation (e.g., C5 or higher spinal cord injury as this could affect the clinical course and cloud interpretation of the ventilator-free day endpoint
9. Lack of availability of Dräger Evita Infinity V500 ventilator as this is the only ventilator capable of delivering sigh breaths as described in the protocol
10. Burns > 40% of body surface area as this could affect the clinical course and cloud interpretation of the endpoints
11. Treating physicians being unwilling to use low VT ventilation strategy when ARDS is diagnosed as low VT ventilation is now considered standard of care for patients with ARDS.
12. Moribund, not expected to survive 24 hours as this could affect the clinical course and cloud interpretation of the endpoints13. Treating physician's decision to use airway pressure release ventilation (APRV).
13. Patient not expected to require mechanical ventilation > 24 hours (e.g., intubated for alcohol intoxication rather than pulmonary problem).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2022-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Albert, MD, Principal Investigator — University of Colorado, Denver
Locations (15):
- United States (15):
  - UCSF Fresno Community Regional Medical Center, Fresno, California
  - University of Southern California (LA County), Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - UC San Diego Medical Center, San Diego, California
  - Christiana Care Health System, Newark, Delaware
  - University of Maryland Medical System Shock Trauma Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Medical Center Brackenridge, Austin, Texas
  - UT Southwestern (Parkland), Dallas, Texas
  - University of Texas Medical School, Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albert RK, Jurkovich GJ, Connett J, Helgeson ES, Keniston A, Voelker H, Lindberg S, Proper JL, Bochicchio G, Stein DM, Cain C, Tesoriero R, Brown CVR, Davis J, Napolitano L, Carver T, Cipolle M, Cardenas L, Minei J, Nirula R, Doucet J, Miller PR, Johnson J, Inaba K, Kao L. Sigh Ventilation in Patients With Trauma: The SiVent Randomized Clinical Trial. JAMA. 2023 Nov 28;330(20):1982-1990. doi: 10.1001/jama.2023.21739. PMID 37877609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in 15 trauma centers in the United States from April, 2016, to September, 2022.
Pre-assignment Details: All analyses were based on the intention-to-treat principle. Participants were included in the primary analysis if primary endpoint data was available (ventilator-free days (VFDs), defined as the number of days of unassisted breathing to day 28 without having to re-institute invasive ventilation).
Period: Overall Study
Arm/Group | Sigh Breaths | Usual Care
Started | 261 | 263
Completed | 259 | 261
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sigh Breaths | Usual Care | Total
Number analyzed (Participants) | 261 | 263 | 524
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 43.7 (19.1) | 44.2 (19.2) | 43.9 (19.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 66 | 130
  Male | 197 | 197 | 394
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 42 | 85
  Not Hispanic or Latino | 218 | 221 | 439
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 55 | 52 | 107
  White | 202 | 203 | 405
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 261 | 263 | 524
Smoking status [Count of Participants; unit: Participants]
  Current/Past | 134 | 103 | 237
  Never | 65 | 80 | 145
  Unknown/Missing | 62 | 80 | 142
Arterial blood gas pH [Mean (Standard Deviation); unit: pH] — Population: Data based on available medical records
  pH
    number analyzed (Participants) | 234 | 243 | 477
    (all) | 7.36 (0.08) | 7.37 (0.08) | 7.36 (0.08)
Arterial blood gas PaCO2 [Mean (Standard Deviation); unit: mmHg] — Population: Data based on available medical records
  mmHg
    number analyzed (Participants) | 234 | 243 | 477
    (all) | 39.1 (7.4) | 38.6 (7.8) | 38.9 (7.6)
Arterial blood gas PaO2 [Mean (Standard Deviation); unit: mmHg] — Population: Data based on available medical records
  mmHg
    number analyzed (Participants) | 234 | 243 | 477
    (all) | 157.4 (84.2) | 152.5 (79.9) | 154.9 (82.0)
Arterial blood gas FIO2 [Mean (Standard Deviation); unit: mmHg] — Population: Data based on available medical records
  mmHg
    number analyzed (Participants) | 230 | 228 | 458
    (all) | 48.2 (18.9) | 47.1 (17.2) | 47.6 (18.1)
P/F ratio [Mean (Standard Deviation); unit: Ratio] — Population: Data based on available medical records
  Ratio
    number analyzed (Participants) | 230 | 228 | 458
    (all) | 347.6 (172.0) | 349.8 (214.0) | 349.2 (193.8)
Hours on ventilator prior to randomization [Mean (Standard Deviation); unit: hours] | 17.1 (5.8) | 17.0 (5.9) | 17.0 (5.8)
Injury Severity Score [Mean (Standard Deviation); unit: units on a scale] — Score range, 0 (no injury) to 75 (not survivable). Population: Data based on available medical records
  units on a scale
    number analyzed (Participants) | 256 | 259 | 515
    (all) | 28.8 (12.9) | 29.9 (11.7) | 29.4 (12.3)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (6.4) | 28.4 (6.5) | 28.5 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-free Days (VFDs)
Description: Ventilator-free days (VFDs), defined as the number of days of unassisted breathing to day 28 without having to re-institute invasive ventilation. Patients who died before day 28 were assigned 0 VFDs as were those transferred to a long-term care facility while ventilated.
Time Frame: 28 days
Population: Analysis based on participants with available follow-up data
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sigh Breaths | Usual Care
Number analyzed (Participants) | 259 | 261
days | 18.4 [7.0 to 25.2] | 16.1 [1.1 to 24.4]

2. Secondary Outcome: All-cause Mortality
Description: All-cause 28 day mortality
Time Frame: 28 days
Population: Analysis population based on those with follow-up data available
Measure: Count of Participants; unit: Participants
Arm/Group | Sigh Breaths | Usual Care
Number analyzed (Participants) | 259 | 261
Participants | 30 | 46

3. Secondary Outcome: ICU-free Days
Description: Number of ICU-free days to day 28 after enrollment
Time Frame: 28 days
Population: Analysis based on participants with available follow-up data
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sigh Breaths | Usual Care
Number analyzed (Participants) | 259 | 261
days | 13.7 [2.0 to 20.6] | 11.9 [0.0 to 20.0]

4. Secondary Outcome: Number of Participants With Complications of Treatment
Description: Specifically the number of participants experiencing pneumothorax, ventilator-associated pneumonia, hypotension requiring pressors, or pneumatoceles.
Time Frame: 28 days
Population: Analysis based on participants with available follow-up data
Measure: Count of Participants; unit: Participants
Arm/Group | Sigh Breaths | Usual Care
Number analyzed (Participants) | 259 | 261
Participants
  Pneumothorax | 18 | 20
  Ventilator-associated pneumonia | 57 | 69
  Hypotension requiring pressors | 127 | 120
  Pneumatocele | 1 | 2

5. Secondary Outcome: Discharge Status
Description: Percentage of patients discharged to extended care facilities, on mechanical ventilation, or to in-patient or home hospice
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sigh Breaths | Usual Care
Number analyzed (Participants) | 261 | 263
Participants | 6 | 5

6. Secondary Outcome: Number of Participants Requiring Oxygen Therapy at Discharge
Description: Number of Participants newly requiring continuous oxygen therapy at discharge.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sigh Breaths | Usual Care
Number analyzed (Participants) | 261 | 263
Participants | 20 | 12

ADVERSE EVENTS:
Time Frame: Participants were followed for 28 days
Description: Events were considered serious if any of the following apply:
  1. Fatal event
  2. Life threatening event
  3. Re-hospitalization
  4. Event likely contributed to prolonging hospitalization
  5. Disabling or incapacitating
  6. Serious laboratory abnormality with clinical symptoms
  Events were detected through responses to routine questionnaires and medical chart review at study visits and also by spontaneous self-report. Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Sigh Breaths | Usual Care
All-Cause Mortality (participants affected / at risk) | 30/259 | 46/261
Serious Adverse Events (participants affected / at risk) | 103/259 | 114/261
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sigh Breaths (N=259) | Usual Care (N=261)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 22 (23)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 20 (22)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 13 (15)
Other Respiratory (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (12)
Infection (Infections and infestations) | 9 (10) | 12 (13)
Stroke (Vascular disorders) | 7 (8) | 7 (9)
Gastrointestinal Bleed (Gastrointestinal disorders) | 6 (7) | 6 (6)
Cardiovascular (Cardiac disorders) | 6 (6) | 6 (6)
Septic Shock (Infections and infestations) | 7 (7) | 3 (4)
Hypotension (Cardiac disorders) | 7 (7) | 0 (0)
Hemorrhagic Shock (Infections and infestations) | 6 (6) | 5 (5)
Brain Injury (Nervous system disorders) | 21 (21) | 31 (31)
Other (General disorders) | 8 (9) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02582957/Prot_SAP_000.pdf